CLINICAL TRIAL: NCT00469339
Title: The Role of Family History and Culture in Communal Coping Within Mexican American Families
Brief Title: Risk Communication Within Mexican-American Families
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907140; 07-HG-N140
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-07-08

CONDITIONS: Breast Cancer; Diabetes; Colon Cancer; Cardiovascular Disease
Keywords: Breast Cancer; Diabetes; Colon Cancer; Cardiovascular Disease; Natural History
MeSH Terms: conditions — Breast Neoplasms; Diabetes Mellitus; Colonic Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort of Mexican-American households: cohort of Mexican-American households
  Interventions: Behavioral: Family Health History

INTERVENTIONS:
Behavioral: Family Health History

SUMMARY:
This study will examine what methods work best for encouraging Mexican-American family members to talk about their risk for diabetes, heart disease, breast cancer and colon cancer. Within the Mexican-American community, the family culture provides an important setting in which individuals interpret and share their health information and formulate strategies to engage in health-promoting behaviors. The information from the study will be used to design risk communication approaches for Mexican-American households.

Members of households with at least three adults 18 to 70 years of age who are part of the existing Mexican-American households recruited by the University of Texas M.D. Anderson Cancer Center may be eligible for this study.

Participants are interviewed about their medical history, family history of disease, health behaviors, beliefs about disease and disease risk, experiences living in the United States, and relationships with family members and close friends. They are then provided information about their family risk for diabetes, heart disease, breast cancer and colon cancer, based on the information they provided in the interview. Two additional interviews are conducted over the telephone that include questions about how the participants communicate with family members about their risk and health behaviors.

DETAILED DESCRIPTION:
The current project aims to understand the mechanisms underlying communications about familial risk for common, complex diseases and the development of strategies by Mexican American families to address this risk. For the Mexican American community, the family culture provides an important setting within which individuals will interpret their health information, share health information, and formulate strategies to engage in health promoting behaviors. This family culture can be defined by the family social structure, the degree of acculturation represented by household members, as well as socio-economic factors. Participants for the current project will be recruited from an ongoing population-based cohort of Mexican American households initiated by the Department of Epidemiology at the University of Texas MD Anderson Cancer Center (UTMDACC). At least three adults, two of which are biological relatives, living within the same residence from 160 multigenerational Mexican American households will participate in this study. Medical risk information (feedback) will be provided to participants based upon family history information that they provide about four complex diseases: diabetes, heart disease, breast cancer and colon cancer. The feedback will be randomized in two ways varying who within the family is provided the feedback (Receiver of the Feedback) and what information is provided (Content of Feedback). The data will allow us to examine whether the family-centered feedback approach (where all participating family members receive feedback), rather than the individual-focused feedback approach (where only one participating family member receives feedback), encourages communications regarding disease risk among family members. The medical risk feedback will also be randomized as to whether they receive disease risk information only (predisposing risk feedback) or disease risk information coupled with personalized recommendations for behavior change to reduce risks (predisposing plus enabling feedback). These data will allow us to examine the impact of the content of risk feedback based on the CDC s family health history tool Family Healthware on beliefs concerning the underlying causes and controllability of common diseases. Cross comparisons between the data obtained from who receives the medical risk information and the content of that information will help in understanding the role of beliefs about disease and communication about family risk for disease in the development of shared perceptions of risk and strategies to adopt health promoting behaviors within the family. The role of the familial and cultural context in the communication and strategy development process will also be investigated.

ELIGIBILITY:
* INCLUSION CRITERIA
* Member household of existing population-based cohort of Mexican-American households recruited by the Department of Epidemiology at UTMDACC. The existing population based cohort consists of self-identified Mexican-Americans living in predominantly Mexican-American neighborhoods in the Houston area. All individuals in the cohort are 18 years of age or older and had to be able to complete a personal interview.
* Household includes at least three adults (18 to 70 years of age) who are willing to participate in the study, where at least two of the household participants are related biologically and represent differing generations, and additionally in which one household participant is a spouse or partner of another household participant.
* Ability for each participating household member to complete one in-home survey instrument via computerized assessment tool or personal interview and to complete two telephone interviews.
* Ability of all household participants to speak either English or Spanish.

EXCLUSION CRITERIA

More than two household members are unable to complete the baseline questionnaire using a computerized assessment tool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican-American households@@@
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2007-04-27

PRIMARY OUTCOMES:
Understand how culture and the familial social system facilitate or impede communications regarding family health history and risk for disease, and the development of strategies to adopt health promoting behaviors. | one survey and two telephone interviews
  Understand how culture and the familial social system facilitate or impede communications regarding family health history and risk for disease, and the development of strategies to adopt health promoting behaviors.
Investigate whether the type of personalized risk feedback (predisposing or predisposing plus enabling) affects family members beliefs about the causes and controllability of disease onset and perceived risk for disease. | one survey and two telephone interviews
  Investigate whether the type of personalized risk feedback (predisposing or predisposing plus enabling) affects family members beliefs about the causes and controllability of disease onset and perceived risk for disease.
Investigate whether shared perceptions of risk and beliefs about disease mediates the relationship between communications about family risk and the development of cooperative strategies to adopt health promoting behaviors within the family. | one survey and two telephone interviews
  Investigate whether shared perceptions of risk and beliefs about disease mediates the relationship between communications about family risk and the development of cooperative strategies to adopt health promoting behaviors within the family.
Examine whether a family-centered feedback approach, as compared to an individual-focused approach, encourages communications regarding family risk and the development of strategies to adopt health promoting behaviors within the household. | one survey and two telephone interviews
  Examine whether a family-centered feedback approach, as compared to an individual-focused approach, encourages communications regarding family risk and the development of strategies to adopt health promoting behaviors within the household.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Glass TA, McAtee MJ. Behavioral science at the crossroads in public health: extending horizons, envisioning the future. Soc Sci Med. 2006 Apr;62(7):1650-71. doi: 10.1016/j.socscimed.2005.08.044. Epub 2005 Sep 29. PMID 16198467
- [Background] Green LW. Public health asks of systems science: to advance our evidence-based practice, can you help us get more practice-based evidence? Am J Public Health. 2006 Mar;96(3):406-9. doi: 10.2105/AJPH.2005.066035. Epub 2006 Jan 31. PMID 16449580
- [Background] Susser M. The tribulations of trials--intervention in communities. Am J Public Health. 1995 Feb;85(2):156-8. doi: 10.2105/ajph.85.2.156. No abstract available. PMID 7856769
- [Derived] Lin J, Marcum CS, Wilkinson AV, Koehly LM. Developing Shared Appraisals of Diabetes Risk Through Family Health History Feedback: The Case of Mexican-Heritage Families. Ann Behav Med. 2018 Feb 17;52(3):262-271. doi: 10.1093/abm/kax037. PMID 29538667